CLINICAL TRIAL: NCT04682613
Title: The Impact of School-Based Programs on the Psychological Health of Children and Youth: The Moderating Role of a Teacher Component and Internet-Delivered Content.
Brief Title: Increasing the Effect of a School-based Prevention Program by Teacher Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel-Hai-College
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Primary Prevention
Keywords: prevention-program; body-image; self-esteem; self-care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Program "young In Favor of Myself", active teachers (Experimental): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The teachers will also participate by delivering planned activities to do with their pupils in addition to each week's topic, parallel to the externally-delivered program. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experimental: Prevention Program "young In Favor of Myself", active teachers
- Prevention Program "young In Favor of Myself", passive teachers (Active Comparator): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The teachers won't participate in the program, they will only be present in the classroom during the externally-delivered program. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experimental: Prevention Program "young In Favor of Myself", no teacher involvement

INTERVENTIONS:
Behavioral: Experimental: Prevention Program "young In Favor of Myself", active teachers — Prevention program: "young In Favor of Myself", with teacher participation
  Arms: Prevention Program "young In Favor of Myself", active teachers
Behavioral: Experimental: Prevention Program "young In Favor of Myself", no teacher involvement — Prevention program: "young In Favor of Myself", without teacher participation
  Arms: Prevention Program "young In Favor of Myself", passive teachers

SUMMARY:
Cluster-Randomized Clinical trial, which includes the development and activation of an intervention program among young adolescents and their teachers. Study hypothesis is that the intervention program will yield improvement in adolescents whose teachers participated in the program, in comparison with the adolescents whose teachers weren't involved in the intervention. Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all student participants in the intervention and in the control group, as well as teachers involved in the program, received information about the program and the study and were asked to provide informed consent.

DETAILED DESCRIPTION:
Early adolescent (10-13 years) is characterized by hormonal changes and accelerated physiological growth. Significant risk factors for the physical and mental health of children and adolescents include, among other things, disordered eating patterns, overweight and reduced physical activity, low self-esteem and negative body image.

"In Favor of Myself" is a preventive intervention program. The program's primary goal is to increase adolescents' self-esteem and to prevent negative self-image and body image, as well as to development media literacy. In this study, the investigators will focus on the "Young In Favor of Myself " program, designed for ages 10-12, grades 5 and 6, and its main goal is the development of self-care behaviors, media literacy, positive self-esteem, and body-image. To increase the effect of "Young In Favor of Myself " program, on the adolescents, the investigators have developed a teacher component as an addition to the school-based intervention, usually delivered by college students. The study will first assess the teachers' influence on the program, and then evaluate the difference in adolescent outcomes from the program with or without this supplement.

Results will be measured using the study questionnaire, to be filled out by the participants (both teachers and adolescents) before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, as well as teachers involved in the program, received information about the program and the study and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Teachers of elementary school classes 10-12-year-old students of participating teachers Participants who filled out the questionnaires before and after the program Participants whose parents signed a letter of informed consent.

Exclusion Criteria:

* Participants who didn't complete the questionnaires at baseline or at least twice.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4, Affects by Media subscale. | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included the Media subscale, including 4 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
  The scale will only be used in the child questionnaire, not in the teacher version.
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
  The scale will only be used in the child questionnaire, not in the teacher version.
Change from Baseline in Body Esteem Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001) The scale will be used in both the child and teacher questionnaire versions.
Change from Baseline in Child- Eating Disorder Examination- Questionnaire (Ch-EDE-Q8) | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Child Eating Disorder Examination- Questionnaire short version (EDE-Q8). The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always. EDE-Q provides assessment of eating disorder psychopathology related to anorexia nervosa (AN), bulimia nervosa (BN), and binge-eating disorder (BED). (Kliem et al, 2016) The scale will only be used in the child questionnaire, not in the teacher version.
Change from Baseline in Advertising Scale | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
  The scale will only be used in the child questionnaire, not in the teacher version.
Change from Baseline in Self-Care behaviors | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the program, measuring a change in scores
  Developed by Prof. Moria Golan and assessed in previous research. Includes 14 items which are rated on a 4-point scale: (1) never, (2) rarely, (3) sometimes, (4) always. Items are summed, and higher scores indicate higher self-care behaviors. This questionnaire was designed to assess self care behaviors in adolescents.
  The scale will only be used in the child questionnaire, not in the teacher version.

SECONDARY OUTCOMES:
Change from Baseline in The Connor-Davidson Resilience Scale (CD-RISC) | Measured three times over six months: at baseline, at program termination (immediately after last session), and three months after the completion of the course, measuring a change in scores
  The CD-RISC is based on Connor and Davidson's operational definition of resilience, which is the ability to "thrive in the face of adversity." The scale includes 25 items, from 5 sub-scales:
  Personal competence, high standards, and tenacity Trust in one's instincts, tolerance of negative affect, and strengthening effects of stress Positive acceptance of change and secure relationships Control Spiritual influences Scoring: Scoring of the scale is based on summing the total of all items, each of which is scored from 0-4. For the CD-RISC-25, the full range is therefore from 0 to 100, with higher scores reflecting greater resilience. (Connor KM, Davidson JRT. Depression and Anxiety 2003; 18: 71-82).
  The scale will only be used in the teacher questionnaire, not in the child version.

CONTACTS AND LOCATIONS:
Overall Officials: Moria Golan, Prof., Principal Investigator — Tel Hai College
Locations (1):
- Tel Hai College, Kiryat Shmona, Upper Galilee, Israel

IPD SHARING:
Plan to Share IPD: No